CLINICAL TRIAL: NCT00030693
Title: Intra-Lesional rF-B7.1 Versus rF-Tricom Vaccine In The Treatment Of Metastatic Cancer
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02455; CPMC-IRB-14535; CDR0000069189 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — rF-B7.1 vaccine

ARMS (2):
- Arm I (recombinant fowlpox-B7.1 vaccine) (Experimental): Patients receive rF-B7.1 vaccine intratumorally on day 1.
  Interventions: Biological: recombinant fowlpox-B7.1 vaccine; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Arm II (recombinant fowlpox-TRICOM vaccine) (Experimental): Patients receive fowlpox-TRICOM vaccine intratumorally on day 1.
  Interventions: Biological: recombinant fowlpox-TRICOM vaccine; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: recombinant fowlpox-B7.1 vaccine — Given intratumorally
  Other Names: rF-B7.1; rF-B7.1 vaccine
  Arms: Arm I (recombinant fowlpox-B7.1 vaccine)
Biological: recombinant fowlpox-TRICOM vaccine — Given intratumorally
  Other Names: rF-TRICOM (B7.1.iCAM1-LFA3-Fowlpox)
  Arms: Arm II (recombinant fowlpox-TRICOM vaccine)
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Randomized phase I trial to compare the effectiveness of two different vaccines given directly into the tumor in treating patients who have metastatic solid tumors. Vaccines may make the body build an immune response to kill tumor cells. Infusing the vaccine directly into a tumor may cause a stronger immune response and kill more tumor cells. It is not yet known which vaccine may be more effective in treating metastatic solid tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine and compare the feasibility and clinical toxicity of administering rF-B7.1 and rF-TRICOM vaccines to patients with accessible cutaneous, subcutaneous, or lymph node metastatic tumors.

II. To determine and compare the feasibility and clinical toxicity of administering rF-B7.1 and rF-TRICOM vaccines to patients with accessible visceral metastatic tumors.

III. To determine the optimal dose of rF-B7.1 and rF-TRICOM vaccine delivered by intra-tumoral injection.

IV. To compare the clinical responses and safety profile of patients with cutaneous tumors and visceral tumors who receive rF-B7.1 vaccine to similar patients receiving rF-TRICOM vaccine.

SECONDARY OBJECTIVES:

I. To establish evidence of host anti-tumor immune reactivity following intra-lesional vaccine administration and compare any differences between rF-B7.1 and rF-TRICOM in patients with cutaneous tumors and visceral tumors.

II. To evaluate the quality of life during vaccine administration.

OUTLINE: This is a randomized study with dose-escalation component. Patients are stratified according to tumor location (cutaneous, subcutaneous, or lymph node metastases vs visceral metastases). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive rF-B7.1 vaccine intratumorally on day 1.

ARM II: Patients receive fowlpox-TRICOM vaccine intratumorally on day 1.

Treatment in both arms repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive additional courses.

Three patients from the cutaneous disease (CD) stratum are treated at low-dose in each treatment arm. If no more than 1 of 6 patients experience dose-limiting toxicity (DLT), then 6 additional CD patients are randomized to high-dose treatment. If no more than 1 of these 6 patients experience DLT, then 12 patients from the visceral disease (VD) stratum are randomized to low-dose treatment. If no more than 2 of 12 VD patients experience DLT, then the next cohort of 12 VD patients is randomized to high-dose treatment. If 3 of the original 12 VD patients experience DLT, then 6 additional VD patients receive low-dose treatment. If no more than 3 of 18 patients experience DLT, then 12 VD patients receive high-dose treatment.

Quality of life is assessed at baseline, monthly during therapy, and then at the end of therapy.

Patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic unresectable solid tumors

  * Cutaneous, subcutaneous, lymph node, or visceral tumors that are accessible to imaging and injections
  * No standard therapy available
* At least 1 unidimensionally measurable lesion

  * At least 20 mm for visceral lesions
  * At least 10 mm for cutaneous, subcutaneous, and nodal lesions
* No untreated or edematous metastatic brain lesions

  * At least 6 weeks since prior surgery and/or radiotherapy for brain metastases and no evidence of disease or edema on CT scan or MRI
* No ascites or pleural effusions
* No leptomeningeal disease
* Performance status - ECOG 0-1
* More than 3 months
* Absolute granulocyte count at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis
* Bilirubin no greater than 1.5 mg/dL*
* SGOT/SGPT no greater than 2 times upper limit of normal (ULN)*
* Alkaline phosphatase no greater than 2 times ULN*
* No elevated PT or PTT
* No cirrhosis
* No active hepatitis
* No hepatic insufficiency
* Creatinine no greater than 2.0 mg/dL
* No renal insufficiency
* No chronic obstructive pulmonary disorder
* No active autoimmune disorders
* No active immunologically mediated disease (e.g., severe psoriasis, colitis, idiopathic thrombocytopenic purpura, multiple sclerosis, connective tissue disease, or active rheumatoid arthritis)
* No significant allergy or hypersensitivity to eggs
* No active seizure disorder
* No active or chronic infections
* No other significant medical disease that would preclude study participation
* No other malignancy within the past 5 years except stage I cervical cancer or basal cell carcinoma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 8 weeks since prior immunotherapy and recovered
* More than 4 weeks since prior chemotherapy and recovered
* At least 4 weeks since prior systemic corticosteroids
* No concurrent corticosteroids
* More than 2 weeks since prior radiotherapy and recovered
* No evidence of bone marrow toxicity from prior radiotherapy
* More than 4 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-12; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Percentages of the DLTEs | 12 weeks
  Will be summarized and compared between arms, doses, and disease groups using Fisher's exact test.

SECONDARY OUTCOMES:
Proportion of patients with any response (CR, PR, or SD) | 12 weeks
  First, the proportion with any response (CR, PR or SD) will be compared to those with no response (PD). Secondly, the proportion of any response (CR, PR or SD) compared to no response (PD) will be compared between the two treatment arms.
Immune response | 12 weeks
  Number of T-cells after treatment compared to those measured at baseline, and difference calculated as after-treatment minus baseline. First comparison includes all subjects who completed treatment. Mean change in T-Cells (final-baseline) tested against 0 with 2-tailed, 1-sample t-test, with alpha=.05. Second analysis compares mean change in T-Cells between arms. Performed as a 2-tailed, 2 independent samples t-test, with alpha=.05. Third comparison is a sub-set analysis of patients with melanoma.
Change in quality of life, assessed using the FACT-G survey of emotional and functional well being | Baseline to 12 weeks
  A mean observed change in the FACT-G score will be tested against 0 (no change) for the group as a whole. Secondly, the change in score will be compared between the two treatment arms. The overall mean change will also be compared to historical controls either from the literature for cancer patients or to the values for non-subject cancer patients receiving other therapies. Comparisons will be by t-test if the sample distribution meets parametric assumptions. If not non-parametric procedures will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Kaufman, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States